CLINICAL TRIAL: NCT07385573
Title: A Single Arm Controlled Trial to Evaluate the Safety and Efficacy of the Long (> 150mm) Passeo-18 Lux Drug-coated Balloon of Teleflex in the Treatment of Subjects With Stenotic, Restenotic or Occlusive Lesions of the Femoropopliteal Artery
Brief Title: Evaluation of the Safety and Efficacy of the Long (> 150mm) Passeo-18 Lux Drug-coated Balloon of Teleflex in the Treatment of Subjects With Stenotic, Restenotic or Occlusive Lesions of the Femoropopliteal Artery
Acronym: LUX-PAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KANDO Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUX-PAD
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Drug Coated Balloon; Peripheral Arterial Disease
Keywords: LUX-PAD; Passeo-18 Lux Long; Passeo-18
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Passeo-18 Lux Arm (Experimental): All trial participants will be treated with the same Passeo-18 Lux drug coated balloon (which comes in different sizes).
  Interventions: Procedure: Percutaneous Transluminal Angioplasty with the use of Passeo-18 Lux DCB

INTERVENTIONS:
Procedure: Percutaneous Transluminal Angioplasty with the use of Passeo-18 Lux DCB — This intervention uses the Passeo-18 Lux paclitaxel-releasing percutaneous transluminal angioplasty (PTA) balloon catheter for the treatment of new or recurring cholesterol-related blockages in the arteries of the lower leg.

SUMMARY:
This clinical trial will evaluate the study device, Passeo®-18 Lux® paclitaxel-releasing percutaneous transluminal angioplasty (PTA) balloon catheter for the treatment of new or recurring cholesterol-related blockages in the arteries of the lower leg.

The device that is used in this trial has been assessed in several previous studies for safety and effectiveness. The device is already approved for use in Europe. It has a "CE mark," which means it meets the European Union's safety, health and performance standards.

This trial is being done to gather additional information on how well the device works and how safe it is when used in everyday medical care with specific attention to the longer lengths of the balloon, as it comes in different sizes.

ELIGIBILITY:
Inclusion Criteria:

1. Lesion(s) in the infrainguinal arteries
2. Reference Vessel Diameter 2-7mm
3. De novo stenotic, restenotic post POBA (the phenomenon where atherosclerotic plaques form in the treated arteries after balloon angioplasty), or occlusive lesion(s)
4. Target lesion must have angiographic evidence of ≥70% stenosis
5. Lesion length ≥ 3cm
6. Successful crossing of the target lesion with the guide wire
7. Successful predilatation, defined as residual stenosis <50% without flow limiting dissection grade D, E or F (Modified Fujihara classification)
8. Rutherford Class 2-5
9. Study participant is able to provide consent and has signed and dated the informed consent form

Exclusion Criteria:

1. Life expectancy ≤ 1 year
2. Study participant is currently participating in another investigational drug or device study that has not reached its primary endpoint yet.
3. Study participant is pregnant or planning to become pregnant during the course of the study.
4. Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion).
5. Prior bypass surgery of target vessel
6. In-stent restenosis
7. Planned major amputation of the target limb
8. Thrombus in the target vessel
9. Known allergy to contrast media that cannot be adequately controlled with premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from Clinically Driven Target Lesion Revascularization (TLR) (Primary Clinical Performance Endpoint) | 12-months post-index procedure
  The primary clinical performance endpoint is freedom from clinically driven target lesion revascularization (TLR) within 12 months post-index procedure.
Freedom from Major Adverse Events (MAE) through 12 months | Through 12 months post-index procedure
  The primary safety endpoint is freedom from major adverse events (MAE), defined as a composite of freedom from device- and procedure-related mortality through 30 days, and freedom from major target limb amputation and clinically driven TLR, within 12 months post-index procedure.

SECONDARY OUTCOMES:
Successful delivery, inflation, deflation, and retrieval of the intact study device during index procedure. | During index procedure
  Device success is defined as successful delivery, balloon inflation, deflation, and retrieval of the intact study device without burst below rated burst pressure.
Restoration of target lesion with ≤30% residual stenosis in final angiogram. | After index procedure
  Procedural success is defined as restoration of the target lesion with ≤30% residual stenosis in the final angiogram.
Number of deaths from any cause (all-cause mortality) at 1, 6, 12, 24, 36, 48, and 60 months | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  All-cause mortality is defined as the total number of deaths from any cause among study participants at each scheduled follow-up time point.
Primary patency of target lesion (freedom from clinically driven target lesion revascularization [CD-TLR] and binary restenosis) | At scheduled follow-up visits: 1, 6, 12, and 24 months
  Primary patency is defined as a composite of freedom from clinically driven target lesion revascularization (CD-TLR) and binary restenosis, where restenosis is defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis as assessed by an independent DUS core lab.
Freedom from Clinically-driven Target Lesion Revascularization (TLR) | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  Clinically driven target lesion revascularization (TLR) is defined as any reintervention performed for ≥50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent clinical symptoms.
Freedom from Clinically-driven Target Vessel Revascularization (TVR) | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  Clinically driven TLR is defined as any reintervention performed for ≥50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent clinical symptoms of the patient.
Freedom from major adverse events (MAE: device- or procedure-related mortality, major target limb amputation, and clinically driven TLR) | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  Major adverse events (MAE) are defined as a composite of freedom from device- or procedure-related mortality through 30 days, freedom from major target limb amputation, and freedom from clinically driven target lesion revascularization (TLR).
Amputation-free survival (AFS: alive without major amputation) | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  Amputation-free survival (AFS) is defined as being alive without major amputation.
Freedom from Major Target Limb Amputation | At scheduled follow-up visits: 1, 6, 12, 24, 36, 48, and 60 months
  Major target limb amputation is defined as any amputation above the ankle in the target limb.
Change from baseline in Rutherford classification at 1, 6, 12, and 24 months | At scheduled follow-up visits: 1, 6, 12, and 24 months
  Change from baseline in Rutherford classification will be assessed to evaluate the severity of ischemia in the lower extremities among study participants.
Change from baseline in EQ-5D quality of life score at 1, 6, 12, and 24 months | At scheduled follow-up visits: 1, 6, 12, and 24 months
  Change from baseline in health-related quality of life, as assessed by the EQ-5D questionnaire, will be evaluated among study participants.
Change from baseline in Walking Impairment Questionnaire (WIQ) score at 1, 6, 12, and 24 months | At scheduled follow-up visits: 1, 6, 12, and 24 months
  Change from baseline in functional limitations, as assessed by the Walking Impairment Questionnaire (WIQ), will be evaluated among study participants with peripheral artery disease (PAD).

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to participant privacy concerns and because data sharing was not included in the informed consent.